CLINICAL TRIAL: NCT04317612
Title: A Randomized, Double-blind, Placebo-controlled Intervention Study to Evaluate the Effect of Nordic Berries on Cognitive Function, Cardiometabolic Risk Markers and Gut Microbiome in Adults With Mild Cognitive Impairment The MINDBERRY Trial
Brief Title: Effect of Nordic Berries on Cognitive Function, Cardiometabolic Risk Markers and Gut Microbiota in Adults With Mild Cognitive Impairment
Acronym: MINDBERRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Berry Lab (Unknown)
Responsible Party: Principal Investigator, Maria Landqvist Waldö, Dr., Region Skane
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Mindberry2020
Record Dates: First submitted 2020-03-04; First posted 2020-03-23 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Cognitive Impairment, Mild; Memory Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active berry product (Active Comparator): Once daily consumption over the period of the study
  Interventions: Other: Active berry product
- Reference product (Placebo Comparator): Once daily consumption over the period of the study
  Interventions: Other: Reference product

INTERVENTIONS:
Other: Active berry product — Subjects should consume the active product containing nordic berries daily during the 12 week intervention period.
  Arms: Active berry product
Other: Reference product — Subjects should consume a reference product (isocaloric to active product) daily during the 12 week intervention period.
  Other Names: inactive control
  Arms: Reference product

SUMMARY:
The aim of the current study is to investigate whether daily intake of Nordic berries for 12 weeks can improve cognitive abilities of adults with mild cognitive impairment, and whether the effect can be linked to changes in metabolic parameters.

DETAILED DESCRIPTION:
The study will be conducted with a randomized, double-blind, parallel-group (2 arms) placebo-controlled, single-center interventional design. The aim is to investigate the effects on cognitive function and cardiometabolic risk markers after 12 weeks intake of a berry product vs. a reference product. The reference will be isocaloric and matched in taste, appearance, volume and macronutrient composition to the active berry product.

Two groups, each of 50 volunteers, are studied. Volunteers will be patients attending the Cognitive medicine unit at Ängelholm hospital, who have mild cognitive impairment (but not dementia). One group of volunteers will consume the berry product while the other group act as control and will consume the reference product.

Each volunteer will be seen for a screening visit as well as one pre- and one post-intervention visit at the clinic. In addition, there will be 2 follow-up calls in between visits. Pre- and post-intervention visits will include cognitive assessment with the CANTAB battery (episodic memory and verbal recognition memory), as well as additional cognitive and behavioral tests. Cardiometabolic parameters will be addressed (plasma glucose, insulin, inflammatory markers, blood lipids, body composition) and fecal samples collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 55 years or older.
2. Cognitive impairment in accordance with the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria and global deterioration scale (GDS) stage 3.
3. Capable and willing to give written informed consent.
4. Capable and willing to perform cognitive testing (mastering the Swedish language, functional vision and hearing or the use of visual or hearing aids during testing).
5. Capable and willing to ingest the study beverage for 12 weeks and to follow the instructions given.

Exclusion Criteria:

1. MMSE (Mini-Mental State Examination) <24 (at screening or in the last 3 months).
2. Cognitive disease (e.g. dementia) according to Global Deterioration Scale (GDS) stage 4 and up.
3. Severe affective disorder with current symptoms
4. Severe mental disorder.
5. Newly diagnosed or poorly regulated thyroid disease (unstable dose since 3 months back).
6. Ongoing insulin therapy.
7. Ongoing treatment for malignancy*.
8. Conditions with major impact on the gastrointestinal tract (such as Crohn's disease, ulcerative colitis, diagnosed gluten intolerance, undertaken intestinal resection or weight loss surgery).
9. Planned major intervention in health care over the next 3 months (the study period).
10. Undergoing antibiotic therapy for the last 3 months prior to inclusion in the study.
11. Allergy / intolerance to berries or other ingredients in the study products (i.e., colorants, aromas, starch).
12. Vegetarians / vegans.
13. Smoking.
14. Abuse of alcohol or psychoactive substance.
15. Significant change in medication over the last 3 months.
16. Daily, regular high consumption of berries or juices / marmalade / product with high content of these berries (guideline no more than 5 grams per day). (Can be recruited for the study if this intake ceases before visit 1. High consumes (approximately 1 dl of berries per day) has to cease with this at least one month before visit 1.)
17. Taking supplements with potential cognitive effects (e.g. omega-3, ginko biloba), or containing grape and berry extracts or probiotics (capsules or other). (Can be recruited if this intake ceases at least one month before visit 1).
18. Planned longer absence/vacation during the next 3 months (the study period).
19. Concurrent participation in other clinical intervention trials (dietary/pharmacological).
20. Other reasons that make the Study investigator in consultation with the responsible physician deem the person inappropriate to include.

    * basalioma exempt from exclusion criteria.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
CANTAB - Paired Associate Learning test (PAL28) | 12 weeks
  To investigate how daily berry intake affects cognitive function (primary objective) measured by episodic memory

SECONDARY OUTCOMES:
Episodic memory (test verbal recognition memory (VRM) (free-, immediate- and delayed recall) | 12 weeks
Attention, psychomotor speed and executive function (Trail making test (TMT) A and B) | 12 weeks
Selective attention and processing speed (Stroop color-word test) | 12 weeks
Verbal fluency (letter "S" word fluency test) | 12 weeks
  Number of novel words on letter "S" during 60 seconds.
Behavior and quality of life (AES, Apathy evaluation score (self)) | 12 weeks
  Answers given by the participants on 18 questions reflect apathy including behavioral, cognitive and emotional indicators on a scale 18-72 where higher scores reflect more apathy.
Behavior and quality of life (Apathy evaluation score (informant)) | 12 weeks
  Answers given by someone close to the participant on 18 questions reflect apathy including behavioral, cognitive and emotional indicators on a scale 18-72 where higher scores reflect more apathy.
EuroQol five dimension (EQ-5D) life quality score. | 12 weeks
  Participant marks on a visual analogue scale from 0 to 100 how they value their current health status where 0 represents the lowest, and 100 highest, health status and quality of life.
Hospital Anxiety Depression (HAD) Score. | 12 weeks
  Self-assessment with 14 items that assess anxiety and depression symptoms before and after the intervention on a scale from 0 to 21, with higher scores indication the presence of symptoms.
Systolic blood pressure | 12 weeks
  Change in systolic blood pressure in mm/Hg
Diastolic blood pressure | 12 weeks
  Change in diastolic blood pressure in mm/Hg
Heart rate | 12 weeks
  Change in bpm (beats per minute)
Body weight | 12 weeks
  Change in body weight (kg)
BMI | 12 weeks
  Change in body weight index (kg/m^2)
Body fat composition | 12 weeks
  Body fat composition (% body fat, fat free mass (kg), basal metabolic rate (BMR) measured with TANITA scale.
Waist-to-hip ratio | 12 weeks
  Waist circumference/hip circumference
Fasting glucose (mM) | 12 weeks
Fasting insulin | 12 weeks
HOMA-IR | 12 weeks
  Homeostasis model assessment of insulin resistance (HOMA-IR)
Lipid metabolism: total cholesterol mg/dl | 12 weeks
Lipid metabolism: LDL-cholesterol mg/dl | 12 weeks
Lipid metabolism: HDL-cholesterol mg/dl | 12 weeks
Lipid metabolism: triglycerides mg/dl | 12 weeks
Lipid metabolism: apolipoprotein B/ apolipoprotein A1 ratio | 12 weeks
Lipid metabolism: oxLDL | 12 weeks
  Oxidized LDL-cholesterol
Liver function: alanine aminotransferase (ALAT) (ukat/L) | 12 weeks
Inflammation: hsCRP (mg/L) | 12 weeks
  high sensitive c-reactive protein
Inflammation: plasma serum amyloid A (mg/L) | 12 weeks
Inflammation: IL-6 ng/L | 12 weeks
Inflammation: TNFalfa ng/L | 12 weeks
Inflammation: IL-12 ng/L | 12 weeks
Inflammation: IL-15 ng/L | 12 weeks
Inflammation: MCP-1 ng/L | 12 weeks
Inflammation: sVCAM-1 (ukat/L) | 12 weeks
Inflammation: IFN-g | 12 weeks
Biomarker related to cognitive function: BDNF | 12 weeks
  Change in plasma brain-derived neurotrophic factor (BDNF)
PAL scores (PALTEA) | 12 weeks
  Change in PALTEA score at different levels of the test
VRM scores | 12 weeks
  Change in VRM scores at different levels of the test

OTHER OUTCOMES:
Gut microbiota composition | 12 weeks
  Change in 16s microbial composition in feces samples
Gut function | 12 weeks
  Questionnaire describing gut function and habits to be filled out before and after the intervention.
Exploratory: correlations between primary variables (cognitive function) and secondary outcome measures and gut microbiota composition. | 12 weeks
Exploratory: analyses of interactions between effects on cognitive function and the participant characteristics; dietary habits, drugs, dementia risk-allele, education level and gender. | 12 weeks
Adverse events | 12 weeks
  safety outcomes

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Cognitve medicine, Ängelholm
  - Cognitive medicine, Ängelholm

IPD SHARING:
Plan to Share IPD: No